CLINICAL TRIAL: NCT02020967
Title: Programme of Acromegaly Screening in Patients With Associated Somatic Disorders, Who Are Observed at the Moscow Board of Health Endocrinology Dispensary and Endocrinology Hospital at First Moscow State Medical University for the Purpose of Early Identification of the Disease.
Brief Title: Programme of Acromegaly Screening in Patients With Associated Somatic Disorders
Acronym: ACROSCREEN
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-52030-280
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Results first posted 2021-04-28 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acromegaly patients
  Interventions: Other: Non-interventional cross-sectional survey

INTERVENTIONS:
Other: Non-interventional cross-sectional survey — This is a survey which does not involve any intervention into routine clinical practice, including the use of any investigational therapy or special examination methods.

SUMMARY:
The primary objective of the protocol is to define percentage of patients with acromegaly in relation to the total number of screened patients with confirmed clinically significant set of associated somatic disorders with the help of laboratory (Insulin-like Growth Factor I, Growth Hormone, Oral Glucose-Tolerance Test [IGF-1, GH, OGTT]) and instrumental examination methods (Magnetic Resonance Imaging [MRI]).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and above with associated somatic disorders observed at the Moscow Endocrinology dispensary or Endocrinology Hospital at First Moscow State Medical University
* Patients who signed the Informed Consent Form for participation in the survey before collection of any information.

Exclusion Criteria:

* Patient already diagnosed with acromegaly
* Patient's refusal to participate in the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with somatic disorders associated with acromegaly, who are observed at the Moscow Board of Health Endocrinology dispensary and Endocrinology Hospital at First Moscow State Medical University
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2013-12-05 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- Russia (2):
  - Moscow Board of Health Endocrinology Dispensary, Moscow
  - Endocrinology Hospital at First Moscow State Medical University, Moscow

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional cross-sectional survey conducted at 2 clinical sites in Russia between 05 December 2013 and 15 September 2015. This survey did not involve any intervention into routine clinical practice, including the use of any investigational therapy or special examination methods.
Pre-assignment Details: Adults with somatic disorders associated with acromegaly who were observed as out-patients were eligible, and 367 participants were enrolled in the survey focused on early acromegaly diagnosis. Participants previously diagnosed with acromegaly were excluded.
Groups:
- All Participants: Participants did not receive any investigational therapy or special examination methods. Participants screening was implemented in the following stages:
  1. Questioning stage: Participant's and Investigator's questionnaires. Based on the outcome of this stage, participants proceeded to the stage of examination to confirm acromegaly using biochemical assays.
  2. Stage of examination: Insulin-like growth factor 1 (IGF-1) level was measured. In case of increased IGF-1 level, growth hormone (GH) test before and after oral glucose tolerance test (OGTT) was conducted. If acromegaly was confirmed, pituitary magnetic resonance imaging (MRI) with contrast was made.
Period: Overall Study
Arm/Group | All Participants
Started | 367
Examined Participants | 329
Completed (Completed Participation in the Survey.) | 316
Not Completed | 51
Not completed — Withdrawal by Subject | 51

BASELINE CHARACTERISTICS:
Population: The Examined population included all participants for whom blood samples were taken for the biochemical assays to diagnose acromegaly.
Groups:
- Acromegaly Diagnosed: Participants did not receive any investigational therapy or special examination methods. Participants were diagnosed with acromegaly by biochemical assays.
- No Acromegaly Diagnosed: Participants did not receive any investigational therapy or special examination methods. Participants were not diagnosed with acromegaly.
- Total: Total of all reporting groups
Arm/Group | Acromegaly Diagnosed | No Acromegaly Diagnosed | Total
Number analyzed (Participants) | 9 | 320 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (8.22) | 58.0 (13.11) | 58.0 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 268 | 275
  Male | 2 | 52 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Diagnosed With Acromegaly
Description: Acromegaly is an acquired pathological condition related to excessive production of growth hormone and characterized by somatic disfigurement and multiple systemic manifestations. The percentage of participants with acromegaly was determined in participants with a confirmed clinically significant set of associated somatic disorders using biochemical assays (IGF-1, GH, OGTT) and instrumental examination methods (MRI).
Time Frame: Participants were screened over approximately 21 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Groups:
- All Participants: Participants did not receive any investigational therapy or special examination methods. Participants screening was implemented in the following stages:
  1. Questioning stage: Participant's and Investigator's questionnaires. Based on the outcome of this stage, participants proceeded to the stage of examination to confirm acromegaly using biochemical assays.
  2. Stage of examination: IGF-1 level was measured. In case of increased IGF-1 level, GH test before and after OGTT was conducted. If acromegaly was confirmed, pituitary MRI with contrast was made.
Arm/Group | All Participants
Number analyzed (Participants) | 329
percentage of participants
  Biochemical assays | 5.8
  Pituitary MRI | 2.4

2. Secondary Outcome: Number of Participants Diagnosed With Acromegaly Using Biochemical Assays (IGF-1, GH, OGTT) and Instrumental Examination Methods (MRI)
Description: Acromegaly is an acquired pathological condition related to excessive production of growth hormone and characterized by somatic disfigurement and multiple systemic manifestations. The number of participants with acromegaly was determined in participants with a confirmed clinically significant set of associated somatic disorders using biochemical assays (IGF-1, GH, OGTT) and instrumental examination methods (MRI).
Time Frame: Participants were screened over approximately 21 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 329
Participants
  Biochemical assays | 19
  Pituitary MRI | 8

3. Secondary Outcome: Percentage of Participants With Associated Concurrent Somatic Disorders
Description: The percentage of participants with associated concurrent somatic disorders were reported in relation to confirmation of acromegaly diagnosis. Concurrent disorders were prior history of condition or diagnosis.
Time Frame: At baseline (Day 1)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Acromegaly Diagnosed | No Acromegaly Diagnosed
Number analyzed (Participants) | 9 | 320
percentage of participants
  Lips enlargement | 22.2 | 3.8
  Typical change of appearance and enlargement of limbs | 100.0 | 56.9
  Headache | 100.0 | 71.9
  Dyspnoea, decrease of working capacity | 55.6 | 80.9

4. Secondary Outcome: Percentage of Participants With Microadenomas and Macroadenomas
Description: Participants were counted as having a microadenomas or macroadenomas if they had at least one microadenoma or macroadenoma during the study. Microadenoma is a benign pituitary tumour size <=10 millimeter (mm) and macroadenoma is a benign pituitary tumour size >10 mm. The percentage of participants with microadenomas and macroadenomas registered during pituitary MRI examination were reported.
Time Frame: Participants were screened over approximately 21 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 329
percentage of participants
  Pituitary MRI performed: Microadenoma (<= 10 mm) | 0.3
  Pituitary MRI performed: Macroadenoma (>10 mm) | 2.1
  Pituitary MRI performed: No adenoma detected | 2.7
  No pituitary MRI performed | 94.8

5. Secondary Outcome: Percentage of Participants With the Most Pathognomonic Subjective and Objective Signs for Tracing Acromegaly
Description: Acromegaly diagnosed based on a clinically significant set of associated somatic disorders and was assessed by logistic regression and canonical discriminant analysis. The likelihood of acromegaly diagnosis, based on a clinically significant set of associated somatic disorders (predictors) was assessed by logistic regression and canonical discriminant analysis. To investigate the extent to which each of the somatic disorders poses a risk factor for acromegaly diagnosis, all predictor variables were entered into each analysis. The percentage of participants predicted to have acromegaly or not is presented for the logistic regression analysis and the canonical discriminant analysis.
Time Frame: Participants were screened over approximately 21 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Acromegaly Diagnosed | No Acromegaly Diagnosed
Number analyzed (Participants) | 9 | 320
percentage of participants
  Logistic regression: Acromegaly | 0 | 0
  Logistic regression: No acromegaly | 2.74 | 97.26
  Canonical discriminant analysis: Acromegaly | 1.52 | 10.94
  Canonical discriminant analysis: No acromegaly | 1.22 | 86.32
Statistical Analysis 1: Comparison: Acromegaly Diagnosed vs No Acromegaly Diagnosed; Predictor variable: Lips enlargement; Test type: Other; p = 0.0196, Regression, Logistic; Odds Ratio (OR) = 7.34, 95% CI 2-sided [1.38 to 39.11]

ADVERSE EVENTS:
Groups:
- All Participants: Participants did not receive any investigational therapy or special examination methods. Participants were involved in the survey focused on early acromegaly diagnosis.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes